CLINICAL TRIAL: NCT01520545
Title: Study to Assess the Safety of 3 mg/mL Gablofen® (Baclofen Injection) Delivered by Intrathecal Administration Using the Synchromed® II Programmable Infusion System
Brief Title: Safety Study of 3 mg/mL Baclofen Injection (Intrathecal) Using A Programmable Pump
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Piramal Critical Care, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNS-GAB101US
Record Dates: First submitted 2012-01-23; First posted 2012-01-30 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Severe Spasticity
Keywords: Gablofen; baclofen injection
MeSH Terms: conditions — Muscle Spasticity | interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gablofen 3 mg/mL (baclofen Injection) (Experimental): 3 mg/mL Gablofen (baclofen Injection)
  Interventions: Drug: Gablofen® 3 mg/mL (baclofen injection); Device: SynchroMed® II Programmable Pump

INTERVENTIONS:
Drug: Gablofen® 3 mg/mL (baclofen injection) — This is a prospective twelve-month Phase IIIb clinical safety trial followed by a 2-year, Phase IV study that will be conducted at clinical trial sites that are experienced with the use of intrathecal baclofen. Patients will be followed for the duration of their treatment with Gablofen® (baclofen injection) 3 mg/mL using the SynchroMed® II Programmable Pump or until the study is terminated.
  Other Names: baclofen injection
Device: SynchroMed® II Programmable Pump — Intrathecal programmable pump

SUMMARY:
Safety study to assess the 3 mg/mL baclofen injection (intrathecal) using a programmable pump

DETAILED DESCRIPTION:
This is a prospective 36-month Phase IIIb/IV clinical safety trial that will be conducted at clinical trial sites that are experienced with the use of intrathecal baclofen. All patients will be entered after signing an IRB approved informed consent. Patients will be followed for the duration of their treatment with Gablofen® (baclofen injection) 3 mg/mL using the SynchroMed® II Programmable Pump or until the study is terminated. Patients will be evaluated for clinical complications associated with the use of intrathecal baclofen that are considered signs and symptoms of an inflammatory granuloma, specifically new radicular pain at the level of the catheter tip, and/or spinal cord compression. An MRI scan with and without infusion will be performed (with consent of the patient) to evaluate the potential presence of an inflammatory granuloma if clinical signs exist. Events that may be related to an inflammatory granuloma will be classified as a definite granuloma, possible granuloma, other catheter related problem (confirmed not caused by a granuloma), or other clinical sequelae caused by the underlying disease or other infusion system related event.

ELIGIBILITY:
Inclusion Criteria:

* 4 years of age or older
* Subjects must be clinically diagnosed with sever spasticity and be receiving intrathecal baclofen
* Subjects must have a SynchroMed® II Pump already implanted
* Current treatment with intrathecal baclofen should be at the 2 mg/mL concentration
* Life expectancy greater than or equal to 12 months
* Signed written informed consent
* Ability and willingness to comply with the study protocol for the duration of the study and with follow-up procedures

Exclusion Criteria:

* History or presence of malignancy, with the exception of adequately treated localized skin cancer (basal cell or squamous cell carcinoma) or carcinoma in-situ of the cervix, which is allowed
* History of any allergic reaction to baclofen
* History of inflammatory granulomas with an intrathecal infusion pump
* Any previous history of neuroleptic malignant syndrome or malignant hyperthermia
* As a result of medical review and physical examination, the Investigator considers the subject unfit for the study

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2012-12; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
The rate of inflammatory granulomas in patients given 3 mg/mL Gablofen® (baclofen injection) 3mg/mL by the intrathecal route of administration. | 36-months
  The rate of inflammatory granulomas in patients given 3 mg/mL Gablofen® (baclofen injection) 3mg/mL by the intrathecal route of administration.

SECONDARY OUTCOMES:
Overall safety of 3 mg/mL Gablofen® (baclofen injection) given by the intrathecal route of administration | 36-months
  Overall safety of 3 mg/mL Gablofen® (baclofen injection) given by the intrathecal route of administration

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Francisco, MD, Principal Investigator — University of Texas
Locations (13):
- United States (13):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University, Loma Linda, California
  - Rehabilitation Medicine Department, University of Miami, Miller School of Medicine, Miami, Florida
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Wayne State University, School of Medicine, Dearborn, Michigan
  - Gillette Children's Specialty Healthcare, Saint Paul, Minnesota
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Department of Pediatrics, Nashville, Tennessee
  - Cook Children's Health Care System, Fort Worth, Texas
  - TIRR Memorial Hermann, Houston, Texas
  - University of Utah, Division of PM&R, Salt Lake City, Utah
  - The Medical College of Wisconsin Department of Physical Medicine and Rehabilitation, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2014-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT01520545/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT01520545/SAP_001.pdf